CLINICAL TRIAL: NCT04508010
Title: Comparison of Interactive Voice Response (IVR) and Computer-assisted Telephone Interview (CATI) Mobile Phone Surveys for Non-communicable Disease Risk Factor Surveillance in Bangladesh
Brief Title: Comparison of IVR and CATI Surveys in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Institute of Epidemiology, Disease Control and Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 00007318 - Bangladesh
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Surveys and Questionnaires; Non Communicable Diseases
Keywords: mobile phone surveys; interactive voice response
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data cleaning and analysis will be conducted by a statistician blinded to the study arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVR survey (Experimental): Participants will receive an IVR survey
  Interventions: Other: IVR
- CATI survey (Experimental): Participants will receive a CATI survey
  Interventions: Other: CATI

INTERVENTIONS:
Other: IVR — Participants will receive an IVR survey
  Arms: IVR survey
Other: CATI — Participants will receive a CATI survey
  Arms: CATI survey

SUMMARY:
This study focuses on mechanisms to adapt the performance of interactive voice response (IVR) and computer assisted telephone interviews (CATI) surveys conducted in low-and middle-income (LMIC) setting (Bangladesh) and evaluates how the two survey modalities (IVR and CATI) affect survey metrics, including response, completion and attrition rates.

DETAILED DESCRIPTION:
Using random digit dialing (RDD) sampling technique, participants will be randomized to one of two arms : 1) IVR or 2) CATI. Participants in the first study arm will receive an IVR survey. Participants in the second study arm will receive a CATI survey. Each questionnaire contains a set of demographic questions and one non-communicable disease (NCD) module (alcohol, or tobacco, or diet, or physical activity, or blood pressure and diabetes). We will examine contact, response, refusal and cooperation rates and demographic representativeness by each study arm.

ELIGIBILITY:
Inclusion Criteria:

* Access to a mobile phone
* Greater or equal to 18 years of age
* In Bangladesh, conversant in Bengali language

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6151 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Cooperation Rate #1 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, cooperation rate is defined as I/(I+P+R) where I is complete interviews, P is partial interviews, and R is refusals and breakoffs
Response Rate #4 | Time Frame: Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, response rate is defined as (I+P)/(I+P+R+eU) where I is complete interviews, P is partial interviews, R is refusals and breakoffs, and eU is the estimated eligible proportion of unknowns

SECONDARY OUTCOMES:
Contact Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, contact rate is defined as (I+P+R)/(I+P+R+eU) where I is complete interviews, P is partial interviews, R is refusals and breakoffs, and eU is the estimated eligible proportion of unknowns
Refusal Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, refusal rate is defined as (R)/(I+P+R+eU) where R is refusals and breakoffs, I is complete interviews, P is partial interviews, and eU is the estimated eligible proportion of unknowns

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Gibson, PhD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health; Iqbal Khan, PhD, Principal Investigator — Institute of Epidemiology, Disease Control and Research
Locations (1):
- Institute of Epidemiology, Disease Control and Research, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pariyo GW, Greenleaf AR, Gibson DG, Ali J, Selig H, Labrique AB, Al Kibria GM, Khan IA, Masanja H, Flora MS, Ahmed S, Hyder AA. Does mobile phone survey method matter? Reliability of computer-assisted telephone interviews and interactive voice response non-communicable diseases risk factor surveys in low and middle income countries. PLoS One. 2019 Apr 10;14(4):e0214450. doi: 10.1371/journal.pone.0214450. eCollection 2019. PMID 30969975
- [Background] Gibson DG, Wosu AC, Pariyo GW, Ahmed S, Ali J, Labrique AB, Khan IA, Rutebemberwa E, Flora MS, Hyder AA. Effect of airtime incentives on response and cooperation rates in non-communicable disease interactive voice response surveys: randomised controlled trials in Bangladesh and Uganda. BMJ Glob Health. 2019 Sep 6;4(5):e001604. doi: 10.1136/bmjgh-2019-001604. eCollection 2019. PMID 31565406
- [Background] Gibson DG, Pereira A, Farrenkopf BA, Labrique AB, Pariyo GW, Hyder AA. Mobile Phone Surveys for Collecting Population-Level Estimates in Low- and Middle-Income Countries: A Literature Review. J Med Internet Res. 2017 May 5;19(5):e139. doi: 10.2196/jmir.7428. PMID 28476725
- [Background] Hyder AA, Wosu AC, Gibson DG, Labrique AB, Ali J, Pariyo GW. Noncommunicable Disease Risk Factors and Mobile Phones: A Proposed Research Agenda. J Med Internet Res. 2017 May 5;19(5):e133. doi: 10.2196/jmir.7246. PMID 28476722